CLINICAL TRIAL: NCT05187819
Title: Accuracy of Blood-based Biomarkers in Diagnosing Alzheimer's Disease in Clinical Practice
Brief Title: Blood-based Biomarkers for Diagnosis of Alzheimer's
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2730
Record Dates: First submitted 2021-12-24; First posted 2022-01-12 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Dementia Alzheimers
Keywords: Alzheimer's dementia; Diagnosis; Biomarkers; Clinical practice
MeSH Terms: conditions — Alzheimer Disease; Disease

STUDY DESIGN:
Intervention Model Description: A blood test will be taken from patients included. All included patients will have possible early dementia symptoms. A random sample of patients with negative and with positive blood-test results for actual biomarkers for Alzheimer's disease will be referred for further investigation at the memory outpatient clinic in Stavanger. The diagnosis from the memory clinic will be compared with the test results for the biomarkers, in order to calculate the positive and negative predictive value for these biomarkers in general practice.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The results of the blood tests will be hidden for all involved until the investigation at the outpatients clinic is finished. Only the researchers will get the answers for the blood tests.
  The researchers will also get the results from investigation at the outpatient clinic, including test results of biomarkers in CSF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with positive blood test for biomarkers for Alzheimer's disease (Experimental): The positive blood tests results for this group will be compared with the results from the investigation at the at the memory outpatient clinic to calculate the number of false positive blood tests (using the results from the outpatient clinic as a "gold standard" for the diagnosis)
  Interventions: Diagnostic Test: predictive value of a blood test
- Patients with negative blood test for biomarkers for Alzheimer's disease (Active Comparator): The negative blood tests results for this group will be compared with the results from the investigation at the at the memory outpatient clinic to calculate the number of false negative blood tests (using the results from the outpatient clinic as a "gold standard" for the diagnosis)
  Interventions: Diagnostic Test: predictive value of a blood test

INTERVENTIONS:
Diagnostic Test: predictive value of a blood test — Evaluation of the clinical value of a new blood based test for diagnosis of Alzheimer's disease in a general practice population.

SUMMARY:
Alzheimer's disease (AD) may currently be diagnosed using molecular biomarkers in cerebrospinal fluid (CSF) and/or positron emission tomography (PET). These diagnostic procedures are highly accurate, but the high cost and low availability hamper their feasibility. Recently, ultrasensitive blood tests predicting Alzheimer pathologies in the brain have been developed. These tests have a reliable ability to differentiate AD from other neurodegenerative disorders and identify AD across the clinical continuum with high sensitivity and specificity in research cohorts with a high prevalence of AD.

This project will assess the predictive value of these tests in a general practice population.

The hypothesis is that the actual blood panel will have high positive predictive value for a diagnosis of Alzheimer's disease in the primary health care setting.

DETAILED DESCRIPTION:
A correct diagnosis of dementia is important in order to provide the patient and relatives with right information, and to give adequate treatment and support, but also to improve research and further development of treatment. Alzheimer's disease (AD) is the cause of nearly 2/3 of cases of dementia. Current diagnostic methods to ensure accurate diagnosis include analysis of cerebrospinal fluid and molecular PET, but these methods are expensive and not widely available.

Progress has been made in the development of blood-based diagnostic biomarkers for Alzheimer's disease. It will lead to significant simplification and improvement of clinical practice if simple blood tests that can be taken in general practice can provide a reliable diagnosis of Alzheimer's disease.

Several biomarkers (including phosphorylated tau 181, phosphorylated tau 217, phosphorylated tau 231, plasma glial fibrillary acidic protein, plasma β-amyloid 42 to β-amyloid 40 ratio, and plasma neurofilament light) has documented to be useful to distinguish Alzheimer's dementia from non-Alzheimer's dementia in research cohorts with a high prevalence of AD. This project aims to analyze the diagnostic ability of such biomarkers in a primary care cohort with a lower prevalence of AD.

The Stavanger region in Norway will be the catchment area for recruitment of study participants. The region is geographically distinct with 373,000 inhabitants, 15 municipalities with 320 GPs in 94 clinics, all served by one hospital. Consequently, the region offers unique opportunities for community-wide implementation research.

All General Practitioners (GPs) in the region will be invited to, upon consent, select participants for the study. To reflect real-life medical practice in primary care, broad inclusion criteria have been chosen. Blood samples will be taken at the GP offices. First, the robustness of the samples regarding temperature, time and transportation to the laboratory will be studied. Second, the results of the blood samples will be compared with the results of standard diagnostic procedures at the memory outpatient clinic at the hospital. A random sample of an equal number of patients with positive and negative blood biomarker test-results will undergo blinded specialist examination, including MRIs of the brain and analysis of the cerebrospinal fluid for Alzheimer biomarkers. The diagnosis made by the specialists will then be compared to the blood-test results in order to estimate the positive and negative predictive value of such biomarkers for the diagnosis of AD in general practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants suspected by their GP to have possible dementia, based on history, clinical examination and/or cognitive screening

Exclusion Criteria:

* Lack of capacity for consent as judged by the GP.
* Severe psychiatric disease, use of medication or physical disease that according to the GP may affect participation or likely contribute significantly to the observed cognitive impairment.
* Patients not wanting to be referred to the memory outpatient clinic.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The positive predictive value | 2 years
  The positive predictive value of the blood biomarkers for diagnosing Alzheimer's disease in general practice
The negative predictive value | 2 years
  The positive predictive value of the blood biomarkers for diagnosing Alzheimer's disease in general practice

CONTACTS AND LOCATIONS:
Overall Officials: Svein Skeie, MD PhD, Study Director — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No